CLINICAL TRIAL: NCT07211711
Title: Treatment of Temporomandibular Joint Disorders With a Stabilizing Occlusal Splint in Somatosensory Tinnitus: a Randomized Double-blind Placebo-controlled Clinical Trial
Brief Title: Treatment of Temporomandibular Joint Disorders With a Stabilizing Occlusal Splint in Somatosensory Tinnitus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Jeanne Oiticica, PhD, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 67418823.4.0000.0068
Record Dates: First submitted 2025-09-02; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Tinnitus; TMJ; Temporomandibular Disorders (TMD)
Keywords: tinnitus; temporomandibular disorders; TMD; temporomandibular joint; TMJ; bite splint; occlusal splint; splint; stabilizing splint; somatosensory tinnitus
MeSH Terms: conditions — Tinnitus; Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients with temporomandibular joint disorder and somatosensory tinnitus using occlusal splint (Active Comparator): They will undergo the use of a stabilizing occlusal splint and will be followed up for 4 months.
  Interventions: Device: Stabilizing occlusal splint
- Patients with temporomandibular joint disorder and somatosensory tinnitus using placebo splint (Placebo Comparator): They will undergo the use of a placebo splint and will be followed up for 4 months.
  Interventions: Device: placebo splint

INTERVENTIONS:
Device: Stabilizing occlusal splint — Maxillary stabilizing occlusal splint, made of acrylic with 2mm thickness in the posterior region. Installed and evaluated monthly for 4 months.
  Arms: Patients with temporomandibular joint disorder and somatosensory tinnitus using occlusal splint
Device: placebo splint — Maxillary placebo non-occlusal splint, installed and evaluated monthly for 4 months.
  Arms: Patients with temporomandibular joint disorder and somatosensory tinnitus using placebo splint

SUMMARY:
This clinical trial aims to investigate whether treatment of temporomandibular joint disorder with a stabilizing occlusal splint is justified to alleviate somatosensory tinnitus. The main questions we aim to answer are:

* Determine if treatment of temporomandibular disorder with a stabilizing occlusal splint improves somatosensory tinnitus.
* Identify which patient-related, tinnitus-related, and temporomandibular disorder-related factors contribute to the therapeutic effect.

DETAILED DESCRIPTION:
The clinical variables of somatosensory tinnitus (ZS) will be assessed by a researcher blinded to the treatment type, using the Tinnitus Handicap Inventory (THI) and Visual Analogue Scale (VAS) at time points T1, T2, T3, T4, and T5, with 30 days interval. The THI, validated and adapted to Portuguese, is the most frequently used questionnaire in clinical trials for tinnitus patients, quantifying the subjective impact of tinnitus on quality of life across three main domains: functional, emotional, and catastrophic. THI classifies tinnitus into five grades: (a) I - negligible (0-16); (b) II - mild (18-36); (c) III - moderate (38-56); (d) IV - severe (58-76); (e) V - catastrophic (78-100). Audiometry and psychoacoustic measures of tinnitus (pitch, loudness, minimum masking level) will be performed at T1 and T5 by an audiologist blind to the treatment group.

The clinical variables of temporomandibular dysfunction (TMD) will also be assessed by a researcher blinded to the treatment type, using the Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) and VAS at the same time points. The DC/TMD is a validated tool, adapted to Portuguese, used in clinical trials that provides a systematic assessment, including a standardized clinical examination and questionnaires. This classification system, based on the biopsychosocial model of pain, includes a physical assessment through Axis I, using reliable and well-operationalized diagnostic criteria, and an assessment of the psychosocial status and pain-related disability through Axis II.

Both assessments will be conducted at T1, T2, T3, T4, and T5.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old;
* Sufferers of somatosensory tinnitus and TMD for more than 6 months;
* Dentition in good health, with at least minimal occlusion up to the second premolars on both sides;
* Availability for at least 4 months of follow-up;
* Able to speak and read the Portuguese language.

Exclusion Criteria:

Pregnant patients; Treatment for TMD in the last 3 months; Treatment for tinnitus in the last 3 months; Use of total or partial removable prostheses Presence of orofacial pain disorders not related to TMD; Medical contraindication to treatment; Reluctance to accept any designated treatment; Unable or unwilling to give informed consent; Language barrier or delay in neuropsychomotor development.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2023-08-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in somatosensory tinnitus after treatment of temporomandibular joint disorder with a stabilizing occlusal splint. | From enrollment to the end of treatment at 4 months
  Tinnitus improvement was monitored using the tinnitus handicap inventory (THI). A 25-item questionnaire measuring tinnitus-related distress. Scores range from 0 to 100. It subjectively quantifies the impact of tinnitus on the patient's quality of life and classifies tinnitus into 5 degrees: I- negligible (0-16); II- mild (18-36); III- moderate (38-56); IV- severe (58-76); V- catastrophic (78-100).

SECONDARY OUTCOMES:
Somatosensory tinnitus distress reduction after treatment of temporomandibular joint dysfunction with a stabilizing occlusal splint. | From enrollment to the end of treatment at 4 months
  Tinnitus distress was monitored by a Visual Analog Scale (VAS): Patients rated tinnitus distress on 10-point scale (0 = none; 10 = extreme)

CONTACTS AND LOCATIONS:
Locations (1):
- University of São Paulo Faculty of Medicine Clinics Hospital, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: ICF